CLINICAL TRIAL: NCT01900938
Title: Comparison Between Continuous Infusion and Intermittent Bolus Injection of Propofol for Deep Sedation During Endoscopic Retrograde Cholangiopancreatography: a Prospective Randomized Controlled Study
Brief Title: Comparison Between Continuous Infusion and Intermittent Bolus Injection of Propofol for Deep Sedation During ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Kyo-Sang Yoo, Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2012-055
Record Dates: First submitted 2013-05-29; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Biliary Tract Diseases; Pancreatic Diseases
Keywords: Cholangiopancreatography; Endoscopic Retrograde
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases | interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent bolus injection of propofol (Active Comparator): A loading dose of 2 mg of midazolam and 0.4 mg/kg of propofol is initially injected and then repeated intermittent bolus injection of 20 mg of propofol is followed according to patients' sedation level.
  Interventions: Procedure: Intermittent bolus injection of propofol; Drug: Midazolam; Drug: Propofol
- Continuous infusion of propofol (Active Comparator): Propofol is continuously administered intravenously via infusion pump starting with 20 mg/kg/hr and then titrated to about 5 mg/kg/hr according to patients' sedation level.
  Interventions: Procedure: Continuous infusion of propofol; Drug: Propofol

INTERVENTIONS:
Procedure: Continuous infusion of propofol — Propofol is continuously administered intravenously via infusion pump starting with 20 mg/kg/hr and then titrated to about 5 mg/kg/hr according to patients' sedation level.
  Arms: Continuous infusion of propofol
Procedure: Intermittent bolus injection of propofol — A loading dose of 2 mg of midazolam and 0.4 mg/kg of propofol is initially injected and then repeated intermittent bolus injection of 20 mg of propofol is followed according to patients' sedation level.
  Arms: Intermittent bolus injection of propofol
Drug: Midazolam
  Arms: Intermittent bolus injection of propofol
Drug: Propofol

SUMMARY:
The aim of this study is to compare sedation efficiency, safety and satisfaction by both endoscopist, assistants, and the patients between continuous infusion and intermittent bolus injection of propofol for deep sedation during ERCP.

DETAILED DESCRIPTION:
The patients undergone ERCP were randomly assigned to either continuous infusion of propofol (continuous group) or midazolam plus intermittent bolus injection of propofol (intermittent group) for deep sedation. In the continuous group, propofol was continuously administered via infusion pump and the doses were determined by sedation assistants monitoring the patients. In the intermittent group, a loading dose of 2 mg of midazolam and 0.4 mg/kg of propofol was initially injected and repeated bolus injection of 20 mg of propofol was followed according to patients' sedation level. Sedation related parameters (total dose of propofol, induction/recovery time, patients' cooperation) and adverse events during the procedure were evaluated. Satisfaction scores by endoscopist, assistant, and patients and difficulty scores of maintaining the sedation by assistants were also graded after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone ERCP for biliary and pancreatic diseases

Exclusion Criteria:

* Comorbid conditions of ASA class 4-5
* Age under 18 years or over 90 years
* Pregnancy
* Past medication history of benzodiazepine or narcotics
* Known allergy to midazolam or propofol
* hypotension (systolic blood pressure <90 mmHg), hypoxemia (SaO2 <90%), or bradycardia (50/min) at baseline measurements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Satisfaction scores by endoscopist | 30 minutes after the procedure

SECONDARY OUTCOMES:
Adverse events for sedation | 1 day after the procedure
Difficulty scores of maintaining the sedation | 30 minutes after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kyo-Sang Yoo, Principal Investigator — Hanyang University Guri Hospital
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea